CLINICAL TRIAL: NCT03924947
Title: A Phase 4 Study to Compare US Marketed Creon Drug Product With Drug Product Manufactured With a Modernized Process at an Alternate Manufacturing Site and With Drug Product Manufactured With the Approved Manufacturing Process at an Alternate Active Pharmaceutical Ingredient Site, in Subjects With EPI Due to Cystic Fibrosis
Brief Title: A Study to Compare US Marketed Creon Manufactured With a Modernized Process at an Alternate Manufacturing Site and Manufactured With the Approved Manufacturing Process at an Alternate Active Pharmaceutical Ingredient Site, in Participants With Exocrine Pancreatic Insufficiency Due to Cystic Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-111; 2017-000578-12 (EudraCT Number)
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Creon; Pancrelipase; ABT-SLV-245; Exocrine Pancreatic Insufficiency (EPI)
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part 1 Double-Blind Creon MP / Creon (Experimental): After receiving open-label currently marketed Creon delayed release (Creon DR) capsules during a pre-randomization period, participants receive double-blind Creon DR capsules manufactured by modernized process pellets (Creon MP) in treatment period 1, followed by double-blind Creon DR capsules in treatment period 2. Participants also receive open-label currently marketed Creon DR for an interval of up to 28 days between periods 1 and 2, and during a 30-day follow-up period after period 2.
  Interventions: Drug: Pancrelipase
- Part 1 Double-Blind Creon / Creon MP (Experimental): After receiving open-label currently marketed Creon DR capsules during a pre-randomization period, participants receive double-blind Creon DR capsules in treatment period 1, followed by double-blind Creon MP in treatment period 2. Participants also receive open-label currently marketed Creon DR for an interval of up to 28 days between periods 1 and 2, and during a 30-day follow-up period after period 2.
  Interventions: Drug: Pancrelipase
- Part 2 Double-Blind Creon AAPIS / Creon (Experimental): After receiving open-label currently marketed Creon DR capsules during a pre-randomization period, participants receive double-blind Creon DR capsules manufactured at an alternate active pharmaceutical ingredient site (Creon AAPIS) in treatment period 1, followed by double-blind Creon DR capsules in treatment period 2. Participants also receive open-label currently marketed Creon DR for an interval of up to 28 days between periods 1 and 2, and during a 30-day follow-up period after period 2.
  Interventions: Drug: Pancrelipase
- Part 2 Double-Blind Creon / Creon AAPIS (Experimental): After receiving open-label currently marketed Creon DR capsules during a pre-randomization period, participants receive double-blind Creon DR capsules in treatment period 1, followed by double-blind Creon AAPIS in treatment period 2. Participants also receive open-label currently marketed Creon DR for an interval of up to 28 days between periods 1 and 2, and during a 30-day follow-up period after period 2.
  Interventions: Drug: Pancrelipase

INTERVENTIONS:
Drug: Pancrelipase — Delayed release capsules
  Other Names: Creon; ABT-SLV-245; Creon MP
  Arms: Part 1 Double-Blind Creon / Creon MP; Part 1 Double-Blind Creon MP / Creon
Drug: Pancrelipase — Delayed release capsules
  Other Names: Creon; ABT-SLV-245; Creon AAPIS
  Arms: Part 2 Double-Blind Creon / Creon AAPIS; Part 2 Double-Blind Creon AAPIS / Creon

SUMMARY:
Part 1 is a study to demonstrate that Creon (pancrelipase) delayed release (DR) capsules manufactured with a modernized process (MP) is non-inferior to currently marketed pancrelipase DR capsules in participants with exocrine pancreatic insufficiency (EPI) due to cystic fibrosis (CF), as measured by coefficient of fat absorption (CFA). Part 2 is a study to demonstrate that Creon (pancrelipase) manufactured with an alternate active pharmaceutical ingredient site (AAPIS) is non-inferior to currently marketed active control (Creon®) in participants with EPI due to CF, as measured by CFA. Safety is evaluated in each part.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a documented diagnosis of Cystic Fibrosis (CF) confirmed by:

  * a sweat chloride test >= 60 mmol/L, and/or
  * documented CF-causing cystic fibrosis transmembrane conductance regulator (CFTR) mutations and clinical features of CF.
* Participant has diagnosis of moderate to severe Exocrine Pancreatic Insufficiency (EPI), as determined by Fecal Elastase 1 (FE-1) < 15 μg/g at screening.
* Participant has EPI that is currently clinically controlled (no clinically overt steatorrhea or diarrhea) under treatment with a commercially available Pancreatic Enzyme Replacement Therapy (PERT), on an individually established dose regimen for more than 3 months prior to Screening, with a daily dose not exceeding 4,000 Lipase Units (LU)/g fat/day or 10,000 LU/kg/day.
* Participant is available for two (if participating in one of the parts) or four (if participating in both parts) hospitalization/confinement periods of 6 to 8 days each during the expected study window.
* Participant is able to consume a diet with 100 g fat/day, a minimum of 1 g/kg of protein/day and normal to low fiber content.

Exclusion Criteria:

* BMI percentile for age less than 10% in participants less than 18 years of age.
* Participant has a history of any of the following gastrointestinal disorders (acute pancreatitis within 6 months prior to Visit 2, chronic pancreatitis, fibrosing colonopathy, distal intestinal obstruction syndrome (DIOS) within 6 months prior to Visit 2, C. difficile infection within 6 months prior to Visit 2, celiac disease, gastric bypass or partial/total gastrectomy, Crohn's disease or other inflammatory bowel disease, small bowel surgery (other than minor resection due to meconium ileus without resultant malabsorption syndrome), or any type of malignancy involving the digestive tract in the last 5 years).
* Participant has a history of any clinically significant endocrine, respiratory (except mild asthma or CF related lung disease), neurological, cardiac, renal, hepatic (including Hepatitis B or C), hematologic or psychiatric disease or disorder, or any other uncontrolled medical illness which might limit participation in or completion of the study.
* Participant requires concomitant treatment with any medication not allowed by the protocol or a prohibited medication is expected to be needed during the study.
* Participant is currently receiving nutritional supplementation via tube feeding (nasogastric, gastrostomy, jejunostomy).
* Participant has clinically significant (as per Investigator's judgment) abnormalities in clinical chemistry, hematology, or urinalysis (excluding findings that are associated with CF) such as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels >= 3 times the upper limit of normal values, or clinically significant (investigator opinion) elevation of uric acid.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (13):
- United States (13):
  - University of Southern California /ID# 164571, Los Angeles, California
  - Landon Pediatric Foundation /ID# 215411, Ventura, California
  - Nemours Children's Health System /ID# 164553, Jacksonville, Florida
  - Central FL Pulmonary Orlando /ID# 164558, Orlando, Florida
  - The Cystic Fibrosis Institute /ID# 210757, Northfield, Illinois
  - University of Iowa Hospitals and Clinics /ID# 164551, Iowa City, Iowa
  - Via Christi Research /ID# 214266, Wichita, Kansas
  - UH Cleveland Medical Center /ID# 206095, Cleveland, Ohio
  - Cleveland Clinic Main Campus /ID# 212853, Cleveland, Ohio
  - Nationwide Children's Hospital /ID# 225628, Columbus, Ohio
  - Children's Hospital of Philadelphia - Main /ID# 208114, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center /ID# 213434, Nashville, Tennessee
  - Virginia Commonwealth University Medical Center Main Hospital /ID# 164574, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 2 independent parts, and gave participants the option to participate in both. The screening period for each Part included an Open Label (OL) Pre-Randomization Period during which participants were expected to receive OL study drug while they were evaluated for eligibility. Therefore, some participants received treatment in the study who were not enrolled per the protocol definition of enrollment (i.e. randomized).
Pre-assignment Details: A total of 36 unique participants enrolled in the study, with 13 participants enrolling in both parts. Participants who decided to participate in Parts 1 or 2 within ≤ 30 days since completion of the other Part did not need to repeat all screening procedures for the second study Part (including the OL Pre-Randomization Period) before beginning in that Part's Double-Blind (DB) Treatment Period.
Groups:
- Part 1 OL Creon: OL currently marketed Creon delayed release (DR) capsules for up to 35 days during a pre-randomization period.
- Part 1 DB Creon MP / Creon: Participants received DB Creon DR capsules manufactured by modernized process (Creon MP) in treatment period 1, followed by DB currently marketed Creon DR capsules in treatment period 2. Participants also received OL currently marketed Creon DR for an interval of up to 28 days between periods 1 and 2, and during a 30-day follow-up period after period 2.
- Part 1 DB Creon / Creon MP: Participants received DB currently marketed Creon DR capsules in treatment period 1, followed by DB Creon MP in treatment period 2. Participants also received OL currently marketed Creon DR for an interval of up to 28 days between periods 1 and 2, and during a 30-day follow-up period after period 2.
- Part 2 OL Creon: OL currently marketed Creon DR capsules for up to 35 days during a pre-randomization period.
- Part 2 DB Creon AAPIS / Creon: Participants received DB Creon DR capsules manufactured at an alternate active pharmaceutical ingredient site (Creon AAPIS) in treatment period 1, followed by DB currently marketed Creon DR Capsules in treatment period 2. Participants also received OL currently marketed Creon DR for an interval of up to 28 days between periods 1 and 2, and during a 30-day follow-up period after period 2.
- Part 2 DB Creon / Creon AAPIS: Participants received DB currently marketed Creon DR capsules in treatment period 1, followed by DB Creon AAPIS in treatment period 2. Participants also received OL currently marketed Creon DR for an interval of up to 28 days between periods 1 and 2, and during a 30-day follow-up period after period 2.
Period: Part 1: Open Label Pre-Randomization
Arm/Group | Part 1 OL Creon | Part 1 DB Creon MP / Creon | Part 1 DB Creon / Creon MP | Part 2 OL Creon | Part 2 DB Creon AAPIS / Creon | Part 2 DB Creon / Creon AAPIS
Started | 26 | 0 | 0 | 0 | 0 | 0
Completed | 26 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Double Blind Period 1
Arm/Group | Part 1 OL Creon | Part 1 DB Creon MP / Creon | Part 1 DB Creon / Creon MP | Part 2 OL Creon | Part 2 DB Creon AAPIS / Creon | Part 2 DB Creon / Creon AAPIS
Started | 0 | 13 | 13 | 0 | 0 | 0
Completed | 0 | 13 | 12 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other, Not Specified | 0 | 0 | 1 | 0 | 0 | 0
Period: Part 1: Double Blind Period 2
Arm/Group | Part 1 OL Creon | Part 1 DB Creon MP / Creon | Part 1 DB Creon / Creon MP | Part 2 OL Creon | Part 2 DB Creon AAPIS / Creon | Part 2 DB Creon / Creon AAPIS
Started | 0 | 13 | 12 | 0 | 0 | 0
Completed | 0 | 13 | 12 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Open Label Pre-Randomization
Arm/Group | Part 1 OL Creon | Part 1 DB Creon MP / Creon | Part 1 DB Creon / Creon MP | Part 2 OL Creon | Part 2 DB Creon AAPIS / Creon | Part 2 DB Creon / Creon AAPIS
Started | 0 | 0 | 0 | 24 (All Part 2 participants with a record of OL Creon in the pre-randomization period; includes 20 randomized participants and 4 screen failures (who received OL Creon in the pre-randomization period but were not randomized). Does not include 3 randomized participants who have no record of OL Creon in the pre-randomization period (note that, per protocol, participants could skip OL pre-randomization period for Part 2 if they started Part 2 within 30 days of the last dose of study drug in Part 1).) | 0 | 0
Completed | 0 | 0 | 0 | 24 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Double Blind Period 1
Arm/Group | Part 1 OL Creon | Part 1 DB Creon MP / Creon | Part 1 DB Creon / Creon MP | Part 2 OL Creon | Part 2 DB Creon AAPIS / Creon | Part 2 DB Creon / Creon AAPIS
Started | 0 | 0 | 0 | 0 | 11 | 12
Completed | 0 | 0 | 0 | 0 | 11 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Double Blind Period 2
Arm/Group | Part 1 OL Creon | Part 1 DB Creon MP / Creon | Part 1 DB Creon / Creon MP | Part 2 OL Creon | Part 2 DB Creon AAPIS / Creon | Part 2 DB Creon / Creon AAPIS
Started | 0 | 0 | 0 | 0 | 11 | 12
Completed | 0 | 0 | 0 | 0 | 11 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population: all randomized participants who started Double-Blind treatment in Parts 1 and 2 (36 unique participants enrolled in the study, with 13 participants enrolling in both parts).
Groups:
- Part 1 DB Creon MP / Creon: Participants received DB Creon MP in treatment period 1, followed by DB currently marketed Creon DR capsules in treatment period 2. Participants also received OL currently marketed Creon DR for an interval of up to 28 days between periods 1 and 2, and during a 30-day follow-up period after period 2.
- Total: Total of all reporting groups
Arm/Group | Part 1 DB Creon MP / Creon | Part 1 DB Creon / Creon MP | Part 2 DB Creon AAPIS / Creon | Part 2 DB Creon / Creon AAPIS | Total
Number analyzed (Participants) | 13 | 13 | 11 | 12 | 49
Age, Customized [Count of Participants; unit: Participants] — Population: Part 1 and Part 2 participants are presented separately.
  Participants
    Part 1: number analyzed (Participants) | 13 | 13 | 0 | 0 | 26
    Part 1: 12 - 18 years | 2 | 1 |  |  | 3
    Part 1: > 18 years | 11 | 12 |  |  | 23
    Part 2: number analyzed (Participants) | 0 | 0 | 11 | 12 | 23
    Part 2: 12 - 18 years |  |  | 1 | 0 | 1
    Part 2: > 18 years |  |  | 10 | 12 | 22
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Part 1 and Part 2 participants are presented separately.
  Participants
    Part 1: number analyzed (Participants) | 13 | 13 | 0 | 0 | 26
    Part 1: Female | 7 | 6 |  |  | 13
    Part 1: Male | 6 | 7 |  |  | 13
    Part 2: number analyzed (Participants) | 0 | 0 | 11 | 12 | 23
    Part 2: Female |  |  | 6 | 3 | 9
    Part 2: Male |  |  | 5 | 9 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Part 1 and Part 2 participants are presented separately.
  Participants
    Part 1: number analyzed (Participants) | 13 | 13 | 0 | 0 | 26
    Part 1: Hispanic or Latino | 1 | 0 |  |  | 1
    Part 1: Not Hispanic or Latino | 12 | 13 |  |  | 25
    Part 1: Unknown or Not Reported | 0 | 0 |  |  | 0
    Part 2: number analyzed (Participants) | 0 | 0 | 11 | 12 | 23
    Part 2: Hispanic or Latino |  |  | 0 | 1 | 1
    Part 2: Not Hispanic or Latino |  |  | 11 | 11 | 22
    Part 2: Unknown or Not Reported |  |  | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Part 1 and Part 2 participants are presented separately.
  Participants
    Part 1: White: number analyzed (Participants) | 13 | 13 | 0 | 0 | 26
    Part 1: White | 13 | 13 |  |  | 26
    Part 2: White: number analyzed (Participants) | 0 | 0 | 11 | 12 | 23
    Part 2: White |  |  | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Part 1 Coefficient of Fat Absorption (CFA)
Description: CFA is calculated as 100*[fat intake - fat excretion]/fat intake. Fat intake was determined from fat content of food consumed on Day 3, 4, 5 of each treatment period. Fat excretion was determined from the content in the stool(s) collected after the first blue dyed stool (exclusive) following administration of the first blue dye marker (day 2) and until the first dyed stool (inclusive) following administration of the second blue dye marker (day 5) during each treatment period.
Time Frame: Up to Day 8 of each DB treatment period
Population: Evaluable Set: participants who completed both treatment periods and had 100% of stool samples collected and analyzed by the laboratory in both treatment periods
Measure: Least Squares Mean (Standard Error); unit: percentage of fat intake absorbed
Groups:
- Part 1 DB Creon: Part 1 participants received DB currently marketed Creon DR capsules in treatment period 1 or 2.
- Part 1 DB Creon MP: Part 1 participants received Creon MP in treatment period 1 or 2.
Arm/Group | Part 1 DB Creon | Part 1 DB Creon MP
Number analyzed (Participants) | 24 | 24
percentage of fat intake absorbed | 85.53 (1.898) | 84.59 (1.898)
Statistical Analysis 1: Comparison: Part 1 DB Creon vs Part 1 DB Creon MP; Double Blind Creon - Double Blind Creon MP; Test type: Non-Inferiority — The pre-specified non-inferiority margin of upper bound of the two-sided 99% confidence interval for the treatment difference was 12%; Least Squares (LS) Mean of Difference = 0.94, 99% CI 2-sided [-2.370 to 4.259], Standard Error of Mean 1.176 — LS mean (standard error [SE]) and LS mean confidence interval (CI) are based on a mixed effects model including sequence, period and regimen as fixed effects and participants within sequence as a random effect

2. Secondary Outcome: Coefficient of Nitrogen Absorption (CNA)
Description: The CNA is calculated as 100*[nitrogen intake - nitrogen excretion]/nitrogen intake. Nitrogen intake was determined from protein content of food consumed on Day 3, 4, 5 of each treatment period. Nitrogen excretion was determined from the content in the stool(s) collected after the first blue dyed stool (exclusive) following administration of the first blue dye marker (day 2) and until the first dyed stool (inclusive) following administration of the second blue dye marker (day 5) during each treatment period.
Time Frame: Up to Day 8 of each DB treatment period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of nitrogen absorbed
Groups:
- Part 1 DB Creon: Part1 participants received currently marketed Creon DR capsules in treatment period 1 or 2.
- Part 2 DB Creon: Part 2 participants received DB currently marketed Creon DR capsules in treatment period 1 or 2.
- Part 2 Double-Blind Creon AAPIS: Participants received Creon DR capsules manufactured at an AAPIS in treatment periods 1 or 2.
Arm/Group | Part 1 DB Creon | Part 1 DB Creon MP | Part 2 DB Creon | Part 2 Double-Blind Creon AAPIS
Number analyzed (Participants) | 24 | 24 | 20 | 20
percentage of nitrogen absorbed | 85.01 (1.058) | 85.04 (1.058) | 85.67 (1.223) | 86.50 (1.223)
Statistical Analysis 1: Comparison: Part 1 DB Creon vs Part 1 DB Creon MP; Creon - Creon MP; Test type: Other — Descriptive; LS Mean of Difference = -0.03, 95% CI 2-sided [-2.456 to 2.392], Standard Error of Mean 1.169 — LS mean (SE) and LS mean CI are based on a mixed effects model including sequence, period and regimen as fixed effects and participants within sequence as a random effect
Statistical Analysis 2: Comparison: Part 2 DB Creon vs Part 2 Double-Blind Creon AAPIS; Creon - Creon AAPIS; Test type: Other — Descriptive; LS Mean of Difference = -0.83, 95% CI 2-sided [-3.005 to 1.345], Standard Error of Mean 1.035 — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Stool Fat
Description: Total amount of fat excreted during the stool collection period. Stool fat was determined from the stool fat in the stool(s) collected after the first blue dyed stool (exclusive) following administration of the first blue dye marker (day 2) and until the first dyed stool (inclusive) following administration of the second blue dye marker (day 5) during each treatment period.
Time Frame: Up to Day 8 of each DB treatment period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: grams
Groups:
- Part 2 DB Creon AAPIS: Part 2 participants received Creon AAPIS in treatment period 1 or 2.
Arm/Group | Part 1 DB Creon | Part 1 DB Creon MP | Part 2 DB Creon | Part 2 DB Creon AAPIS
Number analyzed (Participants) | 24 | 24 | 20 | 20
grams | 44.52 (5.848) | 47.88 (5.848) | 37.46 (4.734) | 34.19 (4.734)
Statistical Analysis 1: Comparison: Part 1 DB Creon vs Part 1 DB Creon MP; Creon - Creon MP; Test type: Other — Descriptive; LS Mean of Difference = -3.36, 95% CI 2-sided [-10.699 to 3.987], Standard Error of Mean 3.541 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Part 2 DB Creon vs Part 2 DB Creon AAPIS; DB Creon - DB Creon AAPIS; Test type: Other — Descriptive; LS Mean of Difference = 3.27, 95% CI 2-sided [-5.172 to 11.702], Standard Error of Mean 4.016 — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Stool Weight
Description: Stool weight was determined from the net weight of the stool samples collected after the first blue dyed stool (exclusive) following administration of the first blue dye marker (day 2) and until the first dyed stool (inclusive) following administration of the second blue dye marker (day 5) during each treatment period.
Time Frame: Up to Day 8 of each DB treatment period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | Part 1 DB Creon | Part 1 DB Creon MP | Part 2 DB Creon | Part 2 DB Creon AAPIS
Number analyzed (Participants) | 24 | 24 | 20 | 20
grams | 861.04 (66.630) | 826.36 (66.630) | 754.91 (87.307) | 771.47 (87.307)
Statistical Analysis 1: Comparison: Part 1 DB Creon vs Part 1 DB Creon MP; Creon - Creon MP; Test type: Other — Descriptive; LS Mean of Difference = 34.68, 95% CI 2-sided [-94.424 to 163.786], Standard Error of Mean 62.253 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Part 2 DB Creon vs Part 2 DB Creon AAPIS; DB Creon - DB Creon AAPIS; Test type: Other — Descriptive; LS Mean of Difference = -16.56, 95% CI 2-sided [-144.418 to 111.298], Standard Error of Mean 60.858 — [estimate comment as in outcome 2, analysis 1]

5. Primary Outcome: Part 2 Coefficient of Fat Absorption (CFA)
Description: as for outcome 1
Time Frame: Up to Day 8 of each DB treatment period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of fat intake absorbed
Arm/Group | Part 2 DB Creon | Part 2 DB Creon AAPIS
Number analyzed (Participants) | 20 | 20
percentage of fat intake absorbed | 87.74 (1.554) | 88.88 (1.554)
Statistical Analysis 1: Comparison: Part 2 DB Creon vs Part 2 DB Creon AAPIS; Double Blind Creon - Double Blind Creon AAPIS; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; LS Mean of Difference = -1.15, 99% CI 2-sided [-4.892 to 2.602], Standard Error of Mean 1.302 — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: overall median 100.0 days. Adverse Events, Part 1 (1st dose through end of given OL or DB period): OL Creon Pre-Randomization: median 32 days; DB Creon: median 6 days; DB Creon MP: median 6 days; OL Creon Post-Randomization: median 53 days. Adverse Events, Part 2 (1st dose through end of given OL or DB period): OL Creon Pre-Randomization: median 26.5 days; DB Creon: median 6 days; DB Creon AAPIS: median 6 days; OL Creon Post-Randomization: median 46 days.
Description: Events during the OL Pre-Randomization Period are reported for the Open Label Safety Analysis Set (participants who received at least 1 dose of OL Creon during any study period). In Part 1, the 31 participants include 5 screen failures who received OL Creon during the pre-randomization period. In Part 2, the 27 participants include 3 randomized participants with no record of OL Creon pre-randomization and 4 screen failures who received OL Creon during the pre-randomization period.
Groups:
- Part 1 OL Creon Pre-Randomization; Part 2 OL Creon Pre-Randomization: OL currently marketed Creon DR capsules for up to 35 days pre-randomization.
- Part 1 DB Creon; Part 2 DB Creon: DB currently marketed Creon DR capsules in treatment period 1 or 2
- Part 1 DB Creon MP: DB Creon MP capsules in treatment period 1 or 2
- Part 1 OL Creon Post-Randomization; Part 2 OL Creon Post-Randomization: OL currently marketed Creon DR capsules post-randomization.
- Part 2 DB Creon AAPIS: DB Creon AAPIS capsules in treatment period 1 or 2
Arm/Group | Part 1 OL Creon Pre-Randomization | Part 1 DB Creon | Part 1 DB Creon MP | Part 1 OL Creon Post-Randomization | Part 2 OL Creon Pre-Randomization | Part 2 DB Creon | Part 2 DB Creon AAPIS | Part 2 OL Creon Post-Randomization
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/26 | 0/25 | 0/26 | 0/27 | 0/23 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/31 | 1/26 | 0/25 | 0/26 | 0/27 | 0/23 | 0/23 | 1/23
Other Adverse Events (participants affected / at risk) | 4/31 | 1/26 | 0/25 | 0/26 | 0/27 | 3/23 | 1/23 | 2/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 OL Creon Pre-Randomization (N=31) | Part 1 DB Creon (N=26) | Part 1 DB Creon MP (N=25) | Part 1 OL Creon Post-Randomization (N=26) | Part 2 OL Creon Pre-Randomization (N=27) | Part 2 DB Creon (N=23) | Part 2 DB Creon AAPIS (N=23) | Part 2 OL Creon Post-Randomization (N=23)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFECTIVE PULMONARY EXACERBATION OF CYSTIC FIBROSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 OL Creon Pre-Randomization (N=31) | Part 1 DB Creon (N=26) | Part 1 DB Creon MP (N=25) | Part 1 OL Creon Post-Randomization (N=26) | Part 2 OL Creon Pre-Randomization (N=27) | Part 2 DB Creon (N=23) | Part 2 DB Creon AAPIS (N=23) | Part 2 OL Creon Post-Randomization (N=23)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT03924947/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT03924947/SAP_001.pdf